CLINICAL TRIAL: NCT02959047
Title: A Double Blind, Randomized Trial of Alirocumab and Plaque Regression in Peripheral Arterial Disease
Brief Title: A Trial of Alirocumab and Plaque Regression in Peripheral Arterial Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Christopher Kramer, Professor, Department of Medicine, Cardiology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19404
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Arterial Disease
Keywords: MRI; PCSK9 inhibition; LDL cholesterol
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — alirocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alirocumab (Experimental): Alirocumab 150mg SQ every 2 weeks
  Interventions: Drug: Alirocumab
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Alirocumab — 150mg SQ every 2 weeks
  Other Names: Praluent
  Arms: Alirocumab
Drug: Matching placebo — SQ every 2 weeks
  Arms: Placebo

SUMMARY:
Peripheral arterial disease (PAD) is characterized by lower limb arterial obstruction due to atherosclerosis. Magnetic resonance imaging (MRI) methods can accurately quantify atherosclerotic plaque in the superficial femoral artery (SFA) in patients with PAD. Such techniques have demonstrated plaque regression with statin therapy over 1 year. Alirocumab is a PCSK9 inhibitor that effectively reduces LDL cholesterol up to 70% in patients on statins or intolerant to statins. The investigators hypothesize that effective low density lipoprotein (LDL) lowering with Alirocumab 150m subcutaneously (SQ) every 2 weeks will regress atherosclerotic plaque in the SFA in patients with PAD over one year compared to placebo. 54 patients with mild-moderate PAD (ankle brachial index or ABI 0.4-0.9) will be randomized to alirocumab 150 mg SQ every 2 weeks or matching placebo at the University of Virginia (UVA) (n=34) and Northwestern (n=20). The primary endpoint is change in atherosclerotic plaque volume in the superficial femoral artery over the 1 year treatment period. Secondary endpoints include changes in peak calf muscle perfusion after thigh cuff occlusion/hyperemia, 6-minute walk distance, and blood biomarkers (LDL cholesterol, fibrinogen, high sensitivity c-reactive protein (hs-CRP), and lipoprotein(a).

DETAILED DESCRIPTION:
PAD is characterized by lower limb arterial obstruction due to atherosclerosis. There are over 8.5 million people with PAD in the U.S. Recent data in a general population over 40 demonstrated an incidence of PAD defined by ankle brachial index (ABI) of 4.3%. Another study of over 3000 patients, mean age 59, demonstrated a prevalence of 3.9%. The prevalence is age-dependent, rising to 14.5% in those over 70. In populations at risk including diabetics or smokers, the incidence is nearly 30%. Standard cardiovascular (CV) risk factors are also risks for PAD, especially smoking, diabetes, hypertension, African-American race and chronic kidney disease. The annual rate of CV events including myocardial infarction, stroke, and CV death is 5-7%. The adjusted risk of dying of a CV event is 2-fold higher than those without PAD.

Magnetic resonance imaging (MRI) methods can accurately quantify atherosclerotic plaque in the superficial femoral artery (SFA) in patients with PAD. These measures can be performed rapidly and reproducibly with an intraclass correlation of 0.997 for intraobserver reproducibility, 0.987 for intraobserver, and 0.996 for test-retest reproducibility, Plaque regression with statins have been shown using these techniques in PAD.

Alirocumab is a PCSK9 inhibitor that effectively reduces LDL cholesterol up to 70% in patients on statins or intolerant to statins. This injectable agent has proven safe and well-tolerated, but has not yet been studied specifically in patients with peripheral arterial disease.The study will be a double blind, placebo-controlled, randomized study of Alirocumab vs. placebo in 54 patients with PAD.

Baseline visit: Informed consent will be signed. Vital signs will be taken and blood drawn fasting for baseline values. A MRI would be performed with black blood imaging of the SFA of both legs. Approximately 10-15 cm of each leg would be covered, using a specifically designed surface coil (Machnet, Leiden, NL). The imaging would start at the bifurcation of the common femoral and proceed distally. The pulse sequence used will be a black blood turbo spin echo proton density weighted sequence with 3mm slice thickness and 3mm gaps that will be subsequently interleaved. A single slice with an extensive amount of plaque will be chosen for imaging of plaque characteristics including T1- and T2-W imaging. Finally, a calf muscle perfusion study will be performed in the leg that is most symptomatic and/or has the lowest ABI in the absence of claudication symptoms. The calf will be wrapped in a flexible surface coil in a 3T scanner. Subjects will be placed supine in the MR scanner with the calf at the magnet isocenter. A thigh cuff will be inflated up to 250 mmHg for 5 min. Arterial spin labeling images of the mid-calf will be obtained immediately after release of the cuff.Regions of interest will be drawn on the relative blood flow maps corresponding to calf muscle groups to measure perfusion in ml/min/100g.

Randomization: The study statistician will do a block randomization and let the pharmacy know. Patients in the treatment group will begin treatment with alirocumab or matching placebo, 150 mg subcutaneously every 2 weeks. Treatment will continue for 26 treatments or 1 year.

Final Visit: This will be a repeat of the initial visit with vital signs, blood draw for lipid panel, and repeat MRI with the exact same protocol as on the initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-85
* Clinical diagnosis of peripheral arterial disease
* Ankle brachial index of 0.4-0.9
* Either on statin for at least 6 months or statin intolerant. The statin used should be a high potency statin (Crestor, Lipitor) or high dose of a lower potency statin (e.g. Zocor 40-80mg, Pravachol 40-80 mg)

Exclusion Criteria:

* rest pain
* critical limb ischemia
* known or planned stent in the SFA
* known occlusion of the SFA
* planned revascularization within the next year
* inability to lie flat
* known contraindications to MRI including pacemaker, implantable cardioverter defibrillators, certain intracranial aneurysm clips, claustrophobia
* pregnancy
* known allergy to alirocumab

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Change in superficial femoral plaque volume (summed from both legs) | 1 year
  Measured by black blood MRI, expressed in cm3

SECONDARY OUTCOMES:
Change in calf muscle perfusion in the most symptomatic leg | 1 year
  Measured by arterial spin labeling MRI, expressed in ml/min/100g
Change in plaque characteristics | 1 year
  % lipid in one slice from each leg
Change in 6-minute walk test | 1 year
  expressed in feet
Change in LDL cholesterol | 1 year
Change in high sensitivity c-reactive protein | 1 year
Change in fibrinogen | 1 year
Change in lipoprotein (a) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Kramer, MD, Principal Investigator — University of Virginia Health System
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rrapo-Kaso E, Loffler AI, Petroni GR, Meyer CH, Walker M, Kay JR, DiMaria JM, Domanchuk K, Carr JC, McDermott MM, Kramer CM. Alirocumab and plaque volume, calf muscle blood flow, and walking performance in peripheral artery disease: A randomized clinical trial. Vasc Med. 2023 Aug;28(4):282-289. doi: 10.1177/1358863X231169324. Epub 2023 Apr 24. PMID 37093712